CLINICAL TRIAL: NCT02308488
Title: PHASE I - II STUDY OF PRONE ACCELERATED BREAST AND NODAL IMRT(Intensity-Modulated Radiation Therapy)
Brief Title: Study of Prone Accelerated Breast And Nodal IMRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0623
Record Dates: First submitted 2014-10-27; First posted 2014-12-04 (Estimated); Results first posted 2022-08-02 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Lymphedema
Keywords: prone IMRT to breast, level III & Supraclavicular; acute toxicity of prone IMRT to breast, level III & SCV
MeSH Terms: conditions — Lymphedema | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Radiation Therapy (Experimental)
  Interventions: Radiation: Intensity-modulated radiation therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy (IMRT) — Patients will receive 15 daily radiation fractions of 2.7 Gy, Monday to Friday for three weeks, to the entire breast/chest wall and axillary level III and supraclavicular nodes with a daily concomitant boost of 0.5 Gy to the tumor bed, for a total daily dose of 3.2 Gy to the tumor bed (2.7 Gy + 0.5 Gy). The overall dose will be 40.5 Gy to the breast/chest wall, axillary level III and supraclavicular nodes, and 48.0 Gy to the tumor bed.

SUMMARY:
Following consent, patients will receive 15 fractions of radiotherapy to the affected breast and to Axillary level III and SCV (Supra-Clavicular) lymph nodes, defined by CT imaging obtained in a prone position using IMRT(intensity modulation radiation therapy ) technique: one fraction daily for 5 days/week for 3 consecutive weeks. Patients will be seen for follow-up at 45-60 days from first radiotherapy treatment, and then yearly. Patients will be assessed for Lymphedema at baseline, end of treatment, and at yearly intervals after completion of radiotherapy. All patients will be followed for toxicity and outcome (local and systemic recurrence, survival). In addition, patients will complete a self-assessment of QOL at baseline, week 3, day 45-60 and 2-yr follow-ups.

DETAILED DESCRIPTION:
A recent Cochrane Collaboration Intervention Review has addressed the effects of altered fractionation size on women with early breast cancer who have undergone breast conservation surgery. Analysis of two prospective randomized trials that included 2644 women, selected based on tumor size less than five cm, negative pathological margin of excision and negative lymph nodes. No difference in clinical outcome was detected. The conclusion of the review is that the use of unconventional fractionation regimens (greater than 2 Gy per fraction) does not affect breast appearance or toxicity, and does not seem to affect local recurrence or five years survival rates.

After breast surgery and an adequate axillary dissection (i.e., at least 8 nodes retrieved in the axillary dissection specimen from level I and II) it is possible to identify patients with 1 - 5 positive nodes who require radiotherapy to both the indexed breast/chest wall and the draining nodal stations that the surgeon did not include in the traditional level I - II axillary dissection, i.e., level III and supraclavicular stations. We are proposing to test a new technique that extends prone set up to also include these lymph node regions. Limiting treatment to the supraclavicular fossa and level III axilla in patients with an adequately dissected axilla is supported by several published studies. Regional nodal recurrences are rare (occurring in 1 - 5%) in patients with early stage invasive breast cancer who have undergone breast conserving therapy. Several institutions choose to treat only the level III axilla and supraclavicular nodal stations in patients who have undergone surgical treatment of level I/II axilla. This technique was documented recently by Liengsawangwong, who utilized CT-delineated nodal stations to improve target coverage of SCV (Supra-Clavicular) and level III axillary nodes in patients who had undergone axillary level I/II dissection and were found to have positive lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Pre- or post-menopausal women with stage II - III breast cancer (AJCC 2002)
* Biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm
* Status post segmental mastectomy or mastectomy and axillary node dissection with removal of at least 8 nodes
* One to 5 involved lymph nodes identified at axillary staging
* At least 2 weeks from last chemotherapy or before chemotherapy
* No more than sixty days from final surgery to simulation if no systemic therapy (includes chemotherapy and Hormonal therapy) is given
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast
* More than 5 involved nodes identified at axillary staging
* Current treatment for active connective tissue disorders, such as lupus or scleroderma
* Pregnant or lactating women
* Less than 35 years old

Ages: 36 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, M.D., Principal Investigator — NYU Laura and Issac Perlmutter Cancer Center
Locations (1):
- Laura and Issac Perlmutter Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 97
Completed | 95
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 95
Age, Continuous [Mean (Full Range); unit: years] | 57.02 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 60
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Toxicity > Grade 2 (Skin Toxicity Grade 3 or Above) Occurring Within 60 Days After First Day of Treatment
Description: "Toxicity Grading per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v 3.0). Please refer to the Protocol Appendix 1 for details.
  Grade 1 - Mild, Grade 2 - Moderate, Grade 3 - Severe, Grade 4 - Life-threatening, Grade 5 - Death"
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 95
Participants | 4

2. Primary Outcome: Number of Participants Who Met Constraints
Description: Treatment feasibility will be evaluated for each participant by the ability to meet all physics dose constraints:
  Target volume dose constraints = PTVTumor: V 48 Gy > 98%, PTVBreast: V 40.5 Gy ≥ 95%. PTVNodesEval: V 38.5 Gy > 95%.
  Normal tissue dose constraints = Heart: V 5 Gy < 5%, Ipsilateral lung: V 10 Gy < 20%, Contralateral lung: V 5 Gy < 15%, Spinal cord: 37.5 Gy maximum, Spinal cord plus 0.5 cm margin: 40 Gy maximum, Thyroid: contralateral lobe 15 Gy maximum, Esophagus: V 30 Gy < 50%, 40.5 Gy maximum, Ipsilateral brachial plexus: 42 Gy maximum, Contralateral breast: Efforts should be made to keep the contralateral breast completely outside the primary beams
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 95
Participants | 95

ADVERSE EVENTS:
Time Frame: 5 years from the first day of treatment
Description: Adverse Events are collected throughout the study period via physical exams, lab assessments as well as patient communications.
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 4/95
Serious Adverse Events (participants affected / at risk) | 1/95
Other Adverse Events (participants affected / at risk) | 87/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=95)
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=95)
Abdominal Bloating (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Altered Mental Status (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Gastrointestinal disorders) | 2
Anxiety (Psychiatric disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 35
Arthritis (Musculoskeletal and connective tissue disorders) | 2
AST elevated (Investigations) | 1
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Atrophy/Symmetry (Skin and subcutaneous tissue disorders) | 31
Autoimmune Thyroiditis (Immune system disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Bone Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bradycardia (Cardiac disorders) | 1
Breast Heaviness (General disorders) | 2
Breast Pain (General disorders) | 26
Bruising on shin (Skin and subcutaneous tissue disorders) | 1
Grease Burn (Injury, poisoning and procedural complications) | 1
Burning urination (Renal and urinary disorders) | 1
Cellulitis (Infections and infestations) | 4
Chest Pain / Tightness (Cardiac disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Chronic Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Creatinine Elevated (Metabolism and nutrition disorders) | 1
Cyst, Upper Back (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cysts, Thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
DCIS, Left (Contralateral) Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decreased Libido (Reproductive system and breast disorders) | 2
Decreased ROM (Musculoskeletal and connective tissue disorders) | 2
Decreased Vision (Eye disorders) | 1
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Dimpling (Skin and subcutaneous tissue disorders) | 9
Diverticulosis (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry Desquamation (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema (Musculoskeletal and connective tissue disorders) | 13
Erythema / Dermatitis (Skin and subcutaneous tissue disorders) | 57
Esophagitis (Gastrointestinal disorders) | 14
Eye Dryness, Left (Eye disorders) | 1
Eyelid Function Disorder (Eye disorders) | 1
Fat Necrosis (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 71
Fever (General disorders) | 3
Fibrosis (Skin and subcutaneous tissue disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Flu Like Sympotms (General disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastroesophageal Reflux (Gastrointestinal disorders) | 2
Generalized Pain (General disorders) | 1
Globus Sensation In Throat (Gastrointestinal disorders) | 1
Goiter (Endocrine disorders) | 1
Headache (Nervous system disorders) | 4
Hematochezia (Gastrointestinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hemorroids (Gastrointestinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hot Flashes (Endocrine disorders) | 57
Hyperglycemia (Endocrine disorders) | 5
Hypernatremia (Investigations) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 18
Hypertension (Cardiac disorders) | 3
Hypothyroidism (Endocrine disorders) | 4
Induration (Skin and subcutaneous tissue disorders) | 3
Infection (Infections and infestations) | 2
Injury (Tore Cartilage) (Injury, poisoning and procedural complications) | 1
Injury-Torn Meniscus Right Knee (Injury, poisoning and procedural complications) | 1
Insomnia (General disorders) | 5
Irritability (Nervous system disorders) | 1
Keratosis (Skin and subcutaneous tissue disorders) | 1
Left Lung Post Radiation changes (General disorders) | 1
Leg Spasms (Nervous system disorders) | 3
Leptomeningeal Disease/ Brain Mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lower Flank Pain (General disorders) | 1
Lymphadema (Blood and lymphatic system disorders) | 10
Mastitis (Infections and infestations) | 1
Memory Impairment (Nervous system disorders) | 2
Moist Desquamation (Skin and subcutaneous tissue disorders) | 2
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Nasal Discharge (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neuralgia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 14
Night Sweats (Endocrine disorders) | 2
Nipple Discharge Left Breast (Reproductive system and breast disorders) | 1
Nipple Inversion (Reproductive system and breast disorders) | 1
Nipple Sensitivity (Skin and subcutaneous tissue disorders) | 2
Nipple, skin fissure (Skin and subcutaneous tissue disorders) | 1
Odynophagia (Gastrointestinal disorders) | 2
Onychomycosis (Infections and infestations) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 9
Palpitations (Cardiac disorders) | 1
Panic Attack-Agoraphobia (Psychiatric disorders) | 1
Paresthesia (Nervous system disorders) | 2
Pathological Fracture R Proximal Femur (Musculoskeletal and connective tissue disorders) | 1
Pleural Effusion, Requiring Vats (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 17
Radiation Folliculitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 11
Rectal Bleeding (Gastrointestinal disorders) | 1
Right Rib Pain On Inspiration And When Coughing (Respiratory, thoracic and mediastinal disorders) | 1
Sensitivity To Cold, Fingers/Toes (Nervous system disorders) | 1
Seroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Sexual/Reproductive Disfunction (Reproductive system and breast disorders) | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Skin Thickening (Skin and subcutaneous tissue disorders) | 14
Sore Throat (General disorders) | 5
Tachycardia (Cardiac disorders) | 1
Telangiectasia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Thromboembolic Event (Blood and lymphatic system disorders) | 2
Thrush (Infections and infestations) | 1
TSH, Elevated (Endocrine disorders) | 1
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary Retention (Renal and urinary disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 3
Uterine Toxicity/Bleeding (Reproductive system and breast disorders) | 1
Vaginal Atrophy/Irritation (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 4
Weight Gain (General disorders) | 1
Weight Loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02308488/Prot_SAP_000.pdf